CLINICAL TRIAL: NCT05915429
Title: Predicting Post-operative Intraocular Lens Tilt Using Optical Coherence Tomography Measurements and Partial Least Squares Regression Modelling
Brief Title: Predicting Lens Tilt Using Optical Coherence Tomography and Partial Least Squares Regression Modelling
Acronym: Tilt
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-004
Record Dates: First submitted 2022-10-05; First posted 2023-06-23 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Cataract
Keywords: IOL; tilt; OCT; Scheimpflug
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Misalignment of IOLs can cause severe loss of visual quality. Different types of misalignment are known. Tilt is one type of misalignment that is thought to play a negative role for the optical performance in eyes with IOL designs, especially, if they have aspheric, toric or multifocal optics.

Due to the fact that tilt has an influence on visual quality, the prediction of the post-operative tilt could improve IOL power calculaton significantly especially for toric IOLs. the Aim of this study is to measure tilt with two modern OCT based devices and one Scheimpflug camera and to predict the post-operative tilt using partial least squares regression.

DETAILED DESCRIPTION:
During cataract surgery an artificial intraocular lens (IOL) is implanted in the eye to replace the lens and to correct the refraction for distance vision. Misalignment of IOLs can cause severe loss of visual quality. Different types of misalignment are known. Tilt, one type of IOL misalignment is thought to play a negative role for the optical performance in eyes with IOL designs, especially, if they have aspheric, toric, or multifocal optics. For example, in the case of aspheric IOLs, it appears that even slight amount of tilt may result not only in the loss of the effect of reducing spherical aberrations but in more severe cases even a worsening of the optical quality compared to spherical IOLs. In the case of toric IOLs, tilt introduces higher order aberrations potentially mimicking astigmatism. In the case of multifocal IOLs, tilt increases higher order aberrations, which leads to decreased visual quality.

Various methods to measure IOL misalignments have been described. Studies assessing the IOL position have used subjective grading methods at the slit lamp examination or a Scheimpflug camera 2 to assess IOL decentration and tilt. The subjective grading at the slitlamp may display considerable variability between examiners. This method is more qualitative than quantitative and does not allow fine resolution when reporting IOL tilt. The fact that the patient has no standardized target to focus on makes the method even less reliable. Scanning methods such as Scheimpflug photos require a very well dilated pupil exceeding 6mm to assess the IOL position. Additionally, it can be difficult to identify the anatomical structures of the eye that need to be used as points of reference. 3 Scheimpflug camera images have been used for assessing IOL tilt previously, but erroneous results, often due to corneal magnification, have diminished their widespread use. Another possibility to assess tilt is the use of Purkinje reflexes. The light reflections of Purkinje images at ocular surfaces to evaluate ocular alignment have recently been utilized. Since light is reflected at all interfaces of media with a difference in refractive index, these reflections, called Purkinje images, can be used to assess tilt and decentration of IOLs. Two different clinically applicable Purkinjemeter system provide the measurement of IOL decentration and tilt. The main problem with Purkinje meters is accessibility, as there are only a few prototypes available worldwide.

The most recently developed method for tilt quantification is the use of optical coherence tomography. This method has several advantages compared to the previous methods: OCT based devices are available in most clinics, the resolution of modern OCT devices is high, and the measurements are reproducible.

Due to the fact that tilt has an influence on visual quality, the prediction of the post-operative tilt could improve IOL power calculation significantly, especially for toric IOLs. In the literature, the prediction of tilt was shown to be acceptable for the orientation of tilt, but not for the amount of tilt. Furthermore, there is disagreement concerning the fact, if the amount of tilt increases or decreases after cataract surgery. Aim of this study is to measure tilt with two modern OCT based devices and one Scheimpflug camera and to predict the post-operative tilt using partial least squares regression. This method was developed by Wold and introduced to ophthalmology previously.

ELIGIBILITY:
Inclusion Criteria:

* planned cataract surgery in one or both eyes
* above 21 years of age

Exclusion Criteria:

* Combined surgery (cataract plus glaucoma/vitreoretinal/corneal surgery)
* Best corrected distance visual acuity below 0.05 Snellen
* Pathologies that could have an influence on the post-operative tilt, such as pseudoexfoliation syndrome or previous ophthalmic trauma, or other reasons for phakodonesis.
* Previous ophthalmic surgery that could have an influence on post-operative tilt such as pars plana vitrectomy
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with planned cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
change of amount of tilt | preoperation visit and 8 weeks postoperation visit
  difference between preoperative amount of tilt in degrees and postoperative tilt in degrees

OTHER OUTCOMES:
change of orientation of tilt in degrees | pre operation visit and 8 weeks post operation visit
  differnece between preoperative orientation of tilt in degrees and postoperative orientation of tilt in degrees
axial eye length | pre operation visit and 8 weeks post operation visit
  axial eye length in mm
anterior chamber depth | pre operation visit and 8 weeks post operation visit
  anterior chamber depth in mm
anterior segment | pre operation visit and 8 weeks post operation visit
  anterior segment (epithelium of the cornea to posterior lens capsule) in mm
lens thickness | pre operation visit and 8 weeks post operation visit
  lens thickness in mm
lens diameter | pre operation visit and 8 weeks post operation visit
  estimated lens diameter in mm
shape factor | pre operation visit and 8 weeks post operation visit
  shape of factor of the lens in mm
corneal radii | pre operation visit and 8 weeks post operation visit
  corneal radii in mm
age | pre operation visit and 8 weeks post operation visit
  age in years

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Principal Investigator — JKU Linz
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria